CLINICAL TRIAL: NCT00835237
Title: Evaluation of GSK Biologicals' Boostrix® Vaccine When Compared With Decavac™ in Adults Aged 65 Years or Older.
Brief Title: Evaluation of GlaxoSmithKline Biologicals' Boostrix® Vaccine in Comparison With Decavac™ Vaccine.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 111413
Record Dates: First submitted 2009-02-02; First posted 2009-02-03 (Estimated); Results first posted 2010-08-05 (Estimated); Last update posted 2020-01-03 (Actual); Status verified 2019-12

CONDITIONS: Tetanus; Acellular Pertussis; Diphtheria; Diphtheria-Tetanus-acellular Pertussis Vaccines
Keywords: Boostrix®; adults
MeSH Terms: conditions — Tetanus; Diphtheria | interventions — Boostrix; Diphtheria-Tetanus Vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Boostrix Group (Experimental): Subjects received a single dose of Boostrix™ (tetanus toxoids, reduced diphtheria toxoids and acellular pertussis vaccine)
  Interventions: Biological: Boostrix®
- Decavac Group (Active Comparator): Subjects received a single dose of Decavac™ (tetanus and diphtheria toxoids vaccine)
  Interventions: Biological: Decavac™

INTERVENTIONS:
Biological: Boostrix® — Intramuscular, single dose.
  Arms: Boostrix Group
Biological: Decavac™ — Intramuscular, single dose.
  Arms: Decavac Group

SUMMARY:
This phase IIIb, observer-blind study will evaluate the immunogenicity and safety of GSK Biologicals' Boostrix® vaccine in adults (extending indication) aged 65 years or older.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes that can and will comply with the requirements of the protocol should be enrolled in the study.
* Males or females 65 years of age and older at the time of study entry.
* Free of an acute aggravation of the health status as established by medical history and medical history and clinical examination before entering into the study.
* Written informed consent from all subjects.

Exclusion Criteria:

* Administration of a diphtheria-tetanus (Td) booster within the previous 5 years.
* Administration of a Tdap vaccine at any time prior to study entry.
* History of diphtheria and/or tetanus and/or pertussis disease.
* Use of any investigational or non-registered drug or vaccine other than the study vaccines within 30 days preceding vaccination, or planned use during the entire study period.
* Administration of other licensed vaccines within 2 weeks (for inactivated vaccines) or 4 weeks (for live vaccines) prior to enrolment in this study, with the exception of influenza, vaccine, which may be administered at any time up to or during the study period, including the day of study vaccination.
* Planned administration of any vaccine not foreseen by the study protocol up to 30 days following vaccination, with the exception of influenza, vaccine, which may be administered at any time up to or during the study period, including the day of study vaccination. Pneumococcal and zoster vaccines can be administered at the discretion of the investigator when the subject comes back at Visit 2.
* Chronic administration of immunosuppressants or other immune-modifying drugs within six months prior to vaccination or planned administration during the study period.
* Any confirmed or suspected immunosuppressive or immunodeficient condition based on medical history and physical examination.
* History of serious allergic reaction following any other tetanus toxoid, diphtheria toxoid or pertussis-containing vaccine or any component of the study vaccines.
* History of encephalopathy within seven days of administration of a previous booster dose of pertussis vaccine that is not attributable to another identifiable cause.
* Progressive neurologic disorder, uncontrolled epilepsy or progressive encephalopathy: pertussis vaccine should not be administered to individuals with these conditions until a treatment regimen has been established and the condition has stabilized.
* Acute (active) clinically significant pulmonary, cardiovascular, hepatic or renal functional abnormality, as determined by clinical evaluation or pre-existing laboratory screening tests.
* Acute disease at the time of vaccination.
* Administration of immunoglobulins and/or any blood products within the three months preceding vaccination, or planned administration during the study period.
* Any medical condition that, in the opinion of the investigator, might interfere with the evaluations required by the study.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 1332 (Actual)
Dates: Start 2009-02-17 (Actual); Primary Completion 2009-07-23 (Actual); Study Completion 2009-10-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (24):
- United States (24):
  - GSK Investigational Site, Tucson, Arizona
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, DeLand, Florida
  - GSK Investigational Site, West Palm Beach, Florida
  - GSK Investigational Site, Stockbridge, Georgia
  - GSK Investigational Site, Indianapolis, Indiana
  - GSK Investigational Site, Pratt, Kansas
  - GSK Investigational Site, Lexington, Kentucky
  - GSK Investigational Site, Metairie, Louisiana
  - GSK Investigational Site, Columbia, Maryland
  - GSK Investigational Site, Elkridge, Maryland
  - GSK Investigational Site, Milford, Massachusetts
  - GSK Investigational Site, Stevensville, Michigan
  - GSK Investigational Site, High Point, North Carolina
  - GSK Investigational Site, Wilmington, North Carolina
  - GSK Investigational Site, Cleveland, Ohio
  - GSK Investigational Site, Mogadore, Ohio
  - GSK Investigational Site, Wadsworth, Ohio
  - GSK Investigational Site, Mt. Pleasant, South Carolina
  - GSK Investigational Site, Bristol, Tennessee
  - GSK Investigational Site, Fort Worth, Texas
  - GSK Investigational Site, West Jordan, Utah
  - GSK Investigational Site, Williamsburg, Virginia
  - GSK Investigational Site, Wenatchee, Washington

IPD SHARING:
Plan to Share IPD: Yes
IPD is available via the Clinical Study Data Request site (click on the link provided below)
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com/Posting.aspx?ID=150

REFERENCES:
- [Background] Weston WM, Friedland LR, Wu X, Howe B. Vaccination of adults 65 years of age and older with tetanus toxoid, reduced diphtheria toxoid and acellular pertussis vaccine (Boostrix((R))): results of two randomized trials. Vaccine. 2012 Feb 21;30(9):1721-8. doi: 10.1016/j.vaccine.2011.12.055. Epub 2011 Dec 31. PMID 22212127
- [Background] Weston WM et al. Vaccination of adults 65 years of age and older with tetanus toxoid, reduced diphtheria toxoid, and acellular pertussis vaccine (Boostrix™): results of a randomized clinical trial. Abstract presented at the 45th National Immunization Conference (NIC). Washington, USA, 28-31 March 2011.
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Individual Participant Data Set: 111413 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 111413 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 111413 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 111413 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 111413 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 111413 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 111413 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Groups:
- Boostrix Group: Subjects received a single dose of Boostrix (tetanus toxoids, reduced diphtheria toxoids and acellular pertussis vaccine)
- Decavac Group: Subjects received a single dose of Decavac (tetanus and diphtheria toxoids vaccine)
Period: Overall Study
Arm/Group | Boostrix Group | Decavac Group
Started | 887 | 445
Completed | 881 | 445
Not Completed | 6 | 0
Not completed — Lost to Follow-up | 4 | 0
Not completed — Withdrawal by Subject | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Boostrix Group | Decavac Group | Total
Number analyzed (Participants) | 887 | 445 | 1332
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.6 (5.35) | 71.9 (5.62) | 71.7 (5.44)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 478 | 237 | 715
  Male | 409 | 208 | 617

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Antibody Concentration Against Vaccine Antigens, Above a Protocol Defined Cut-off Value
Description: Antibodies against vaccine antigens assessed were: anti-diphtheria (anti-D) and anti-tetanus (anti-T).
  Anti-D antibody cut-off value assessed was ≥ 0.1 International Unit per milliliter (IU/mL)
  Anti-T antibody cut-off values assessed were ≥ 0.1 IU/mL and ≥ 1.0 IU/mL
Time Frame: One month after vaccination.
Population: Analysis was performed on the According-To-Protocol (ATP) cohort for analysis of immunogenicity, on subjects with available results
Measure: Number; unit: subjects
Arm/Group | Boostrix Group | Decavac Group
Number analyzed (Participants) | 864 | 439
subjects
  Anti-D (≥ 0.1 IU/mL) (N= 859;432) | 729 | 374
  Anti-T (≥ 0.1 IU/mL) (N= 864;439) | 836 | 428
  Anti-T (≥ 1.0 IU/mL) (N= 864;439) | 767 | 395

2. Primary Outcome: Anti-pertussis Toxoid (PT), Anti-filamentous Haemagglutinin (FHA) and Anti-pertactin (PRN) Antibodies Concentration
Description: Concentration for anti-PT, anti-FHA and anti-PRN antibodies given as geometric mean concentration (GMC) in Enzyme-Linked Immuno Sorbent Assay (ELISA) units per millilitre (EL.U/mL)
Time Frame: Before (PRE) and one month after vaccination (POST)
Population: Analysis was performed on the ATP cohort for analysis of immunogenicity, on subjects with available results
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | Boostrix Group | Decavac Group
Number analyzed (Participants) | 865 | 439
EL.U/mL
  Anti-PT (PRE) (N=859;433) | 6.6 [6.1 to 7.1] | 6.5 [5.8 to 7.2]
  Anti-PT (POST) (N=852;431) | 49.1 [44.9 to 53.7] | 6.4 [5.8 to 7.1]
  Anti-FHA (PRE) (N=848;430) | 50.2 [46.2 to 54.5] | 44.3 [39.5 to 49.5]
  Anti-FHA (POST) (N=835;428) | 689.0 [638.8 to 743.1] | 44.4 [39.7 to 49.7]
  Anti-PRN (PRE) (N=864;439) | 8.1 [7.4 to 8.8] | 7.8 [6.9 to 8.8]
  Anti-PRN (POST) (N=865;439) | 104.2 [91.3 to 118.9] | 7.7 [6.8 to 8.7]

3. Secondary Outcome: Anti-T and Anti-D Antibody Concentrations
Description: Concentrations for anti-T and anti-D antibodies given as GMC in IU/mL.
Time Frame: Before (PRE) and one month after vaccination (POST)
Population: Analysis was performed on the ATP cohort for analysis of immunogenicity, on subjects with available results
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | Boostrix Group | Decavac Group
Number analyzed (Participants) | 864 | 439
IU/mL
  Anti-D (PRE) (N=844;430) | 0.2 [0.2 to 0.2] | 0.2 [0.1 to 0.2]
  Anti-D (POST) (N=859;432) | 0.9 [0.8 to 1.0] | 0.8 [0.7 to 1.0]
  Anti-T (PRE) (N=864;439) | 0.6 [0.6 to 0.7] | 0.6 [0.5 to 0.7]
  Anti-T (POST) (N=864;439) | 4.0 [3.6 to 4.3] | 7.1 [6.1 to 8.1]

4. Secondary Outcome: Number of Subjects With Vaccine Response for Anti-T and Anti-D Antibodies Concentrations Above the Cut-off
Description: Booster response defined as :
  For initially seronegative subjects (< 0.1 IU/mL), antibody concentration ≥ 0.4 IU/mL one month after vaccination.
  For initially seropositive subjects (≥ 0.1 IU/mL): antibody concentration one month after vaccination ≥ 4 fold the pre-vaccination antibody concentration.
Time Frame: One month after vaccination
Population: Analysis was performed on the ATP cohort for analysis of immunogenicity, on subjects with available results
Measure: Number; unit: subjects
Arm/Group | Boostrix Group | Decavac Group
Number analyzed (Participants) | 863 | 439
subjects
  Anti-D (N=842;428) | 383 | 189
  Anti-T (N=863;439) | 438 | 306

5. Secondary Outcome: Number of Subjects With Vaccine Response for Anti-PT, Anti-FHA and Anti-PRN Antibodies Concentrations Above the Cut-off
Description: Booster response defined as :
  For initially seronegative subjects (< 5 EL.U/mL), antibody concentration ≥ 20 EL.U/mL one month after vaccination.
  For initially seropositive subjects (≥ 5 EL.U/mL) with pre-vaccination antibody concentration < 20 EL.U/mL: antibody concentration one month after vaccination ≥ 4 fold the pre-vaccination antibody concentration.
  For initially seropositive subjects (≥ 5 EL.U/mL) with pre-vaccination antibody concentration ≥ 20 EL.U/mL : antibody concentration one month after vaccination ≥ 2 fold the pre-vaccination antibody concentration.
Time Frame: One month after vaccination
Population: Analysis was performed on the ATP cohort for analysis of immunogenicity, on subjects with available results
Measure: Number; unit: subjects
Arm/Group | Boostrix Group | Decavac Group
Number analyzed (Participants) | 864 | 439
subjects
  Anti-PT (N=846;430) | 585 | 430
  Anti-FHA (N=821;422) | 762 | 7
  Anti-PRN (N=864;439) | 638 | 9

6. Secondary Outcome: Number of Subjects With Vaccine Response for Anti-PT, Anti-FHA and Anti-PRN Antibodies Concentrations Above the Cut-off, Using Alternative Definitions.
Description: Vaccine response using alternative definitions defined as:
  For initially seronegative subjects (< 5 EL.U/mL ), antibody concentration ≥ 10 EL.U/mL one month after vaccination.
  For initially seropositive subjects (≥ 5 EL.U/mL), antibody concentration one month after vaccination ≥ 2 fold the pre-vaccination antibody concentration.
Time Frame: One month after vaccination
Population: Analysis was performed on the ATP cohort for analysis of immunogenicity, on subjects with available results
Measure: Number; unit: subjects
Arm/Group | Boostrix Group | Decavac Group
Number analyzed (Participants) | 864 | 439
subjects
  Anti-PT (N=846;430) | 699 | 9
  Anti-FHA (N=821;422) | 765 | 8
  Anti-PRN (N=864;439) | 714 | 11

7. Secondary Outcome: Number of Subjects Reporting Solicited Local Symptoms
Description: Solicited local symptoms assessed include pain, redness and swelling.
Time Frame: Within the 4-day (Day 0-3) post-vaccination period
Population: Analysis was performed on the Total Vaccinated cohort on subjects with available results
Measure: Number; unit: subjects
Arm/Group | Boostrix Group | Decavac Group
Number analyzed (Participants) | 882 | 445
subjects
  Pain | 190 | 123
  Redness | 95 | 56
  Swelling | 66 | 52

8. Secondary Outcome: Number of Subjects Reporting Solicited General Symptoms
Description: Solicited general symptoms assessed include fatigue, gastrointestinal symptoms, headache, and fever
Time Frame: Within the 4-day (Day 0-3) post-vaccination period
Population: Analysis was performed on the Total Vaccinated cohort on subjects with available results
Measure: Number; unit: subjects
Arm/Group | Boostrix Group | Decavac Group
Number analyzed (Participants) | 882 | 445
subjects
  Fatigue | 110 | 66
  Gastrointestinal symptoms | 67 | 41
  Headache | 101 | 52
  Fever | 18 | 11

9. Secondary Outcome: Number of Subjects Reporting Unsolicited Adverse Events (AE)
Description: An AE is any untoward medical occurrence in a clinical investigation subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.
Time Frame: Within the 31-day (Day 0-30) post-vaccination period
Measure: Number; unit: subjects
Arm/Group | Boostrix Group | Decavac Group
Number analyzed (Participants) | 887 | 445
subjects | 152 | 64

10. Secondary Outcome: Number of Subjects Reporting Serious Adverse Events (SAE)
Description: An SAE is any untoward medical occurrence that: results in death, is lifethreatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect in the offspring of a study subject, or may evolve into one of the outcomes listed above.
Time Frame: From the vaccination up to Day 182
Measure: Number; unit: subjects
Arm/Group | Boostrix Group | Decavac Group
Number analyzed (Participants) | 887 | 445
subjects | 37 | 10

ADVERSE EVENTS:
Arm/Group | Boostrix Group | Decavac Group
Serious Adverse Events (participants affected / at risk) | 37/887 | 10/445
Other Adverse Events (participants affected / at risk) | 351/887 | 202/445
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Boostrix Group (N=887) | Decavac Group (N=445)
Coronary artery disease (Cardiac disorders) | 3 | 0
Myocardial infarction (Cardiac disorders) | 2 | 1
Cerebrovascular accident (Nervous system disorders) | 2 | 0
Hip fracture (Injury, poisoning and procedural complications) | 2 | 0
Pneumonia (Infections and infestations) | 2 | 0
Transient ischaemic attack (Nervous system disorders) | 2 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Angina pectoris (Cardiac disorders) | 1 | 0
Aortic stenosis (Vascular disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Asthenia (General disorders) | 1 | 0
Atrial tachycardia (Cardiac disorders) | 1 | 0
Atrioventricular block complete (Cardiac disorders) | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bone neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Breast cancer in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Carotid artery occlusion (Nervous system disorders) | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 1 | 0
Cervical myelopathy (Nervous system disorders) | 1 | 0
Chest pain (General disorders) | 1 | 0
Complicated migraine (Nervous system disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0
Dementia (Nervous system disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Enterococcal sepsis (Infections and infestations) | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Hernia obstructive (General disorders) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1
Inguinal hernia, obstructive (Gastrointestinal disorders) | 1 | 0
Klebsiella bacteraemia (Infections and infestations) | 1 | 0
Lobar pneumonia (Infections and infestations) | 0 | 1
Meniscus lesion (Injury, poisoning and procedural complications) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 1
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Non-small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteomyelitis (Infections and infestations) | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0
Sick sinus syndrome (Cardiac disorders) | 1 | 0
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Vascular graft occlusion (Injury, poisoning and procedural complications) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Boostrix Group (N=887) | Decavac Group (N=445)
Pain (General disorders) | 190 | 123
Redness (General disorders) | 95 | 56
Swelling (General disorders) | 66 | 52
Fatigue (General disorders) | 110 | 66
Gastrointestinal symptoms (General disorders) | 67 | 41
Headache (General disorders) | 101 | 52

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.